CLINICAL TRIAL: NCT04734678
Title: Comparison of Tocilizumab Versus Tocilizumab/Infliximab in Patients With COVID-19-associated Cytokine Storm Syndrome
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Collaborators: Misr International University (Other)
Responsible Party: Principal Investigator, Neven Sarhan, Lecturer at Faculty of Pharmacy, Misr International University
Other Study IDs: COVID-Infliximab
Record Dates: First submitted 2021-01-31; First posted 2021-02-02 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Covid19; Cytokine Storm; Corona Virus Infection
Keywords: COVID-19; Cytokine Storm; Tocilizumab; Infliximab
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome; Coronavirus Infections | interventions — tocilizumab; Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Moderate and severe patients who were infected with SARS-CoV-2 and received treatment with tocilizumab in addition to standard management.
  Interventions: Drug: Tocilizumab
- Group 2: Moderate and severe patients who were infected with SARS-CoV-2 and received treatment with infliximab and tocilizumab in addition to standard management.
  Interventions: Drug: Tocilizumab; Drug: Infliximab

INTERVENTIONS:
Drug: Tocilizumab — 400 mg IV only once
  Other Names: Actemra
Drug: Infliximab — 5 mg/kg/day IV for 2 doses 12-24 hours
  Other Names: Remicade
  Groups: Group 2

SUMMARY:
Since the end of 2019, Egypt and the whole world have been suffering from the Coronavirus Disease 2019 (COVID-19) pandemic, which is caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). According to the World Health Organization (WHO), since the emergence of this new pandemic, there have been more than 97 million confirmed cases of COVID-19 patients and two million death globally; around 160 thousand of these cases are in Egypt.

Tocilizumab play role among the unique therapeutic alternatives for the management of cytokine release syndrome (CRS), a life-threatening complication of chimeric antigen receptor (CAR) - T cell therapy. CRS occurs as a result of uncontrolled immune activation with release of pro-inflammatory cytokines and chemokines. Up till now, clinical trial and expertise with tocilizumab in COVID-19 patients has been limited. Despite preliminary encouraging results, recent studies suffered from limitations such as the absence of consistent treatment outline, a short post-treatment follow-up, and the absence of a comparison group.

A recent study discussed the possible beneficial effect of tumor necrosis factor (TNF) inhibitors in severe COVID-19. Specifically, TNF may aggravate lymphopenia through direct killing via TNF/TNFR1 signaling in T cells, and T cell dysfunction reveals an important yet underestimated target for immunomodulatory therapeutic approaches. Accordingly, anti-TNF may be considered as an encouraging therapeutic option in severe COVID-19.

These promising clinical findings encouraged us to use infliximab (IFX), a chimeric monoclonal anti-TNF antibody, as an experimental therapy in patients with moderate and severe COVID-19 in the absence of IBD.

In this study, we compare the outcomes of a large cohort of patients with moderate and severe COVID-19 pneumonia treated with tocilizumab in addition to standard management, with those of concomitantly hospitalized patients who received infliximab and tocilizumab in addition to standard management.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years.
2. Able to provide informed consent.
3. Patients hospitalized with pneumonia proved by chest X-ray or CT scan.
4. Confirmed infection with COVID-2019 using RT-PCR or strongly suspected to be infected with pending confirmation studies.
5. Hyper-inflammation defined as elevation in either C-reactive protein (CRP, ≥ 100 mg/L, normal values <6 mg/L) or ferritin (≥ 900 ng/mL, normal value <400 ng/mL), in the presence of increased lactate dehydrogenase (LDH, >220 U/L).
6. And at least one of the following:

   1. Respiratory frequency ≥30/min.
   2. Blood oxygen saturation ≤93% on room air (RA).
   3. Partial pressure of arterial oxygen to fraction of inspired oxygen ratio (PaO2/FiO2) <300 [18].
   4. Worsening of lung involvement, defined as an increase in number and/or extension of pulmonary areas of consolidation, need for increased FiO2 to maintain stable O2 saturation, or worsening O2 saturation of >3% with stable FiO2.

Exclusion Criteria:

1. Evidence of concomitant bacterial infection.
2. Concomitant use of other immunosuppressive biologic drugs.
3. Baseline elevation of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels > 5-fold the upper limit of the normal range.
4. Pregnancy.
5. Treatment with any TNFα inhibitor in the past 30 days.
6. Known hypersensitivity to any TNFα inhibitor, murine proteins, or any component of the formulation.
7. Known or suspected active tuberculosis (TB) or a history of incompletely treated or latent TB.
8. Serious co-morbidity, including:

   1. Myocardial infarction (within last month).
   2. Moderate or severe heart failure (New York Heart Association (NYHA) class III or IV).
   3. Hepatic patients child Pugh class C.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients received the same background treatment for 5 days, following an Institutional protocol for standard of care: hydroxychloroquine 400 mg daily, lopinavir/ritonavir 400/100 mg twice daily or/and remdisivir 200 mg LD then 100 once daily as a maintenance dose and anti-coagulation prophylaxis with enoxaparin subcutaneously once a day if D-dimmer between 500-1000 or enoxaparin therapeutic subcutaneously twice daily if D-dimmer >1000.
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Patients' clinical status improvement using six category scale | Two weeks
  The categories were defined as follows: 1) patient discharged, 2) hospitalization not requiring supplemental oxygen, 3) hospitalization requiring supplemental low-flow oxygen, 4) hospitalization requiring high-flow supplemental oxygen, 5) hospitalization requiring invasive mechanical ventilation, 6) death.
Time to improvement in oxygenation | 48 hours
  Increase in SpO2/FiO2 of 50 or greater compared to the baseline SpO2/FiO2
Duration of hospitalization | Two weeks
  Total admission period
Mortality rate | Two weeks
  Death during hospitalization

SECONDARY OUTCOMES:
Incidence of non-invasive mechanical ventilation | Two weeks
  Need for non-invasive mechanical ventilation
Duration of non-invasive mechanical ventilation | Two weeks
  Time required for non-invasive mechanical ventilation
Incidence of invasive mechanical ventilation | Two weeks
  Need for invasive mechanical ventilation
Duration of invasive mechanical ventilation | Two weeks
  Time required for invasive mechanical ventilation
Occurrence of Secondary infections | Two weeks
  Especially Sepsis
Monitoring of adverse events | Two weeks
  Monitoring of adverse events especially elevation of liver enzymes daily
Occurrence of cardiovascular events | Two weeks
  Prevalence of heart failure, tachycardia and hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Neven Sarhan, PhD, Principal Investigator — Misr International University
Locations (1):
- Teachers Hospital, Cairo, Please Select, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarhan NM, Warda AEA, Ibrahim HSG, Schaalan MF, Fathy SM. Evaluation of infliximab/tocilizumab versus tocilizumab among COVID-19 patients with cytokine storm syndrome. Sci Rep. 2023 Apr 20;13(1):6456. doi: 10.1038/s41598-023-33484-6. PMID 37081046